CLINICAL TRIAL: NCT03718364
Title: Swiss Atrial Fibrillation Pulmonary Vein Isolation Registry
Acronym: SWISS-AF-PVI)
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00226; me18Kuehne2
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Catheter-based Ablation of Atrial Fibrillation
Keywords: atrial fibrillation; pulmonary vein isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During the catheter-based ablation clinically indicated blood samples are necessary to monitor anticoagulation. The excess blood from these analyses and a small amount of blood (50ml per patient) will be stored at -80 C° for future scientific analyses in a central biobank for long term storage. All biobank issues will be handled in accordance with the guidelines published by the Swiss Academy of Medical Sciences (published on www.samw.ch).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: catheter-based ablation of atrial fibrillation (pulmonary vein isolation) — catheter-based ablation of atrial fibrillation (pulmonary vein isolation)

SUMMARY:
Registry of patients with atrial fibrillation undergoing catheter-based ablation of atrial fibrillation (pulmonary vein isolation) to determine long-term success rates of catheter-based ablation of atrial fibrillation (pulmonary vein isolation) and to evaluate factors associated with long-term success of catheter-based ablation of atrial fibrillation (pulmonary vein isolation).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing catheter-based ablation of atrial fibrillation (pulmonary vein isolation)

Exclusion Criteria:

* Patients not able or willing to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing catheter-based ablation of atrial fibrillation (pulmonary vein isolation) at the hospital. The projected duration of the study is open-end with no projected date of study end. Approximately 150-200 patients per year will be included.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2010-07-01 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
changes in retention rate of normal sinus rhythm after catheter-based ablation of atrial fibrillation (pulmonary vein isolation) | before catheter-based ablation of atrial fibrillation and 3, 6 and 12 months after catheter-based ablation of atrial fibrillation
  changes in retention rate of normal sinus rhythm after catheter-based ablation of atrial fibrillation (pulmonary vein isolation)

SECONDARY OUTCOMES:
morphologic changes of left cardiac atrium | before catheter-based ablation of atrial fibrillation (pulmonary vein isolation)
  echocardiography of left cardiac atrium
changes in retention rate of normal sinus rhythm after catheter-based ablation of atrial fibrillation (pulmonary vein isolation) | 12 months after catheter-based ablation of atrial fibrillation and then at intervals of one year until 2035
  changes in retention rate of normal sinus rhythm after catheter-based ablation of atrial fibrillation (pulmonary vein isolation)

OTHER OUTCOMES:
determination of factors associated with long-term success rates of catheter-based ablation of atrial fibrillation | Blood samples gained during catheter-based ablation of atrial fibrillation (pulmonary vein isolation)
  Blood samples (biobanking) for determination of factors associated with long-term success rates of catheter-based ablation of atrial fibrillation (pulmonary vein isolation). Decisions about future analyses to be performed from stored samples will be based exclusively on scientific reasons.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kuehne, MD, Principal Investigator — Cardiology/Electrophysiology, University Hospital Basel
Locations (2):
- Switzerland (2):
  - Cardiology/Electrophysiology, University Hospital Basel, Basel
  - University Hospital Bern, Bern

REFERENCES:
- [Derived] Hennings E, Aeschbacher S, Coslovsky M, Paladini RE, Meyre PB, Voellmin G, Blum L, Kastner P, Ziegler A, Conen D, Zuern CS, Krisai P, Badertscher P, Sticherling C, Osswald S, Knecht S, Kuhne M. Association of bone morphogenetic protein 10 and recurrent atrial fibrillation after catheter ablation. Europace. 2023 Jun 2;25(6):euad149. doi: 10.1093/europace/euad149. PMID 37314197
- [Derived] Meyre PB, Sticherling C, Spies F, Aeschbacher S, Blum S, Voellmin G, Madaffari A, Conen D, Osswald S, Kuhne M, Knecht S. C-reactive protein for prediction of atrial fibrillation recurrence after catheter ablation. BMC Cardiovasc Disord. 2020 Sep 29;20(1):427. doi: 10.1186/s12872-020-01711-x. PMID 32993521